CLINICAL TRIAL: NCT05936814
Title: The Adductor Ratio is More Reliable Than Other Techniques in Determining Joint Line in Severe Type M Varus Gonarthrosis
Brief Title: Adductor Ratio in Severe Varus Gonarthrosis
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, İsmail Demirkale, Clinical professor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Other Study IDs: E-86241737-100--79819
Record Dates: First submitted 2023-06-20; First posted 2023-07-10 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Osteoarthritis, Knee; Genu Varum; Joint Prosthesis; Complications
Keywords: Varus deformity; Adductor tubercle; Joint line restoration; Total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Genu Varum | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intraarticular: The control group with intraarticular varus deformity and Kellgren and Lawrence grade 4 gonarthrosis.
  Interventions: Procedure: total knee arthroplasty
- Metaphyseal: The case group with Metaphyseal varus deformity and Kellgren and Lawrence grade 4 gonarthrosis.
  Interventions: Procedure: total knee arthroplasty

INTERVENTIONS:
Procedure: total knee arthroplasty — cemented bicondylar PCL substituting total knee replacement

SUMMARY:
The restoration of the joint line (JL) is essential for the proper functioning of Total Knee Arthroplasty (TKA). The exact position of JL can be determined using anatomical landmarks such as femoral condylar width (TEW), tibial tubercle, fibular head, and adductor tubercle during preoperative planning or intraoperatively. However, in cases of severe varus deformity in Type M gonarthrosis, it is unknown which method is most suitable for accurately determining the precise JL position. The aim of this study is to identify the most appropriate method for determining the JL position in Type M gonarthrosis. To achieve this goal, two groups of patients with Type 1A and Type M gonarthrosis will be compared by measuring preoperative values and comparing them with intraoperative reference values.

DETAILED DESCRIPTION:
Osteoarthritis (OA) of the knee, known as gonarthrosis, causes significant movement restrictions and pain in daily life activities. Total Knee Arthroplasty (TKA) is the preferred treatment method for advanced-stage OA of the knee. While various alignment techniques such as kinematic, constrained kinematic, and anatomical alignment are used, the most commonly used and preferred method by researchers is TKA performed with a technique that conforms to mechanical alignment.

Two main factors that affect patient outcomes after mechanically aligned TKA are achieving a parallel joint line and appropriate positioning of the distal femoral rotation that corresponds to the patellofemoral joint kinematics, ensuring optimal soft tissue tension. If these two aspects are not adequately addressed, patients may experience chronic pain, functional impairment, early wear at the implant interface, and ultimately, loosening. Studies have reported that 8% to 19% of patients are dissatisfied with TKA due to various reasons, including pain and unmet expectations. Problems that may arise from malrotation and/or incorrect soft tissue tension include patellofemoral instability, anterior knee pain, arthrofibrosis, and flexion gap instability.

In general, the natural joint line is not orthogonal to the tibial mechanical axis; it is varus, ranging from 87 ± 3°. When the mechanical alignment technique is applied in TKA, the proximal tibia and femur are typically cut perpendicular (90°) to the tibial and femoral mechanical axes. However, in the case of symmetric implants, the classical resection technique, especially in varus knees, results in more resection than the component thickness in the medial femoral compartment and the lateral tibial compartment. This creates an average 3° valgus joint line with respect to the tibial mechanical axis. As a result, the joint line is preserved medially, but the lateral compartment becomes more distalized.

Another issue regarding the joint line is its restoration, which involves achieving its anatomical height. Changes in the joint line can lead to instability, increased incidence of anterior knee pain, and decreased range of motion. The most commonly used bone markers for the restoration of the joint line are the epicondyles, fibular head (FH), and tibial tubercle (TT). Due to significant individual variations, some authors have suggested using the ratio of the distance between the epicondyles and the tangent to the joint line to the trans-epicondylar width (TEW) of the femur as a means of determining the appropriate value. This ratio based on femoral width allows for the calculation of an appropriate value for each individual regardless of size. However, it is not always easy to radiographically identify the epicondyles, especially in varus knees with severe metaphyseal damage.

On the femoral side, the width of the distal femoral resection should be equal to the thickness of the metal implant to restore the normal femoral joint line level, regardless of surgical techniques such as "measured resection technique" or modified "gap balancing technique." During surgery, the distal surface of the medial femoral condyle usually serves as the anatomical reference point for the distal femoral cut because in most cases, thicker bone is cut and removed from the medial femoral condyle compared to the lateral condyle. However, in patients with severely degenerated knees, significant bone and cartilage defects occur in the distal femoral condyle, and the deformed medial condyle is no longer a suitable reference point for distal femoral resection.

During total knee arthroplasty (TKA), bone defects are sometimes encountered. If there is insufficient contact between the implant surface and the bone, augmentation is performed on the bone defect to maintain implant stability. Researchers have investigated the use of metal blocks in tibial bone defects during primary TKA and reported positive results, emphasizing that the use of metal blocks is a simple and applicable method for tibial bone defects.

In primary TKA, tibial or femoral defects, or both, are classified into three types by the Anderson Orthopedic Research Institute: Type 1, small defects that do not compromise component stability; Type 2, sponge-like bone loss requiring reconstruction, categorized as A: involving one condyle or B: involving both condyles; Type 3, significant bone loss jeopardizing a large portion of the condyle. Typically, in varus knee deformity, bone defects in the knee appear first in the posteromedial region. In valgus gonarthrosis, the tibial bone defect is central, while the femoral condyles have defects in the distal and posterior lateral regions. Therefore, the primary classification of bone defects includes distinguishing between central forms (defects confined within the peripheral bone cortex) and peripheral forms (characterized by involvement of the peripheral cortex). Additionally, in patients with varus alignment and gonarthrosis, differentiating between intra-articular and metaphyseal sources of alignment defects is crucial as it can lead to differences in postoperative clinical and radiological outcomes, requiring different total knee arthroplasty procedures for patients.

Medial and lateral epicondylar axis (EA) has been used to determine the appropriate location of the joint line (JL) during complex primary total knee arthroplasty (TKA) or most revision TKAs. However, some studies have shown that selecting the epicondyles as a reference can yield significantly different results. In these studies, the maximum errors in intraoperative selection of the medial femoral epicondyle and lateral femoral epicondyle were found to be 7.6 mm and 4.2 mm, respectively. Furthermore, the selection of the medial epicondyle reported more varied results with errors up to 22.3 mm, while the selection of the lateral epicondyle reported errors up to 13.8 mm. Additionally, variations in the distance from the femoral epicondyle to the joint line can be up to 11 mm, and significant differences have been observed between male and female patients. In a study conducted in the researcher's country, a correlation between the adductor tubercle (AT) and the distance between the fibular head (FH) and the JL was investigated to eliminate this handicap and determine the JL instead of using a mathematical ratio between the epicondylar axis and the TEW. The study, conducted on a Turkish population consisting of healthy volunteers, found the average TEW to be 87.2 ± 10.8 mm, the average distance between AT and JL to be 47.9 ± 6.2 mm, and the average distance between FH and JL to be 20.5 ± 4.0 mm. A strong positive correlation (0.55) was found between AT-JL and TEW (adductor ratio - AR). Measurements related to AR calculation were performed on radiographs of young patient knees without osteoarthritis. Based on this, another study questioned the validity of AR by determining the differences between AR in knees with severe osteoarthritis and those without osteoarthritis, considering the significant bone and cartilage loss or osteophyte formation. In revision total knee arthroplasty cases, intraoperative measurement of TEW and calculation of AT-JL may provide more accuracy in determining the articular level compared to measurements taken on radiographs of knees with severe osteoarthritis. They claimed that it could be more logical to measure TEW intraoperatively instead of measuring it on primary or contralateral radiographs of arthritic patients.

According to these two studies, the adductor tubercle can be used as a reliable marker to determine the JL level in complex primary TKA or revision knee arthroplasty surgeries. However, this new method has not been scientifically proven. In fact, there is no generally accepted standard anatomical measurement system to accurately determine the JL level on direct radiographs, especially in severely deformed knees with advanced varus. There is also no consensus on the radiographic appearance to be used and the evaluation of these images. A study found no significant difference (0.01 ± 0.03) between the calculated AR (AT-EA/TEW) ratios obtained from radiographic and intraoperative measurements. This method can be particularly beneficial in revision TKAs where the anatomical EA is not clearly visible and provides a new tool for precise positioning of prosthetic components and JL restoration even in such complex cases.

Literature lacks studies on determining the epicondylar axis using these methods for advanced-stage gonarthrosis cases (Type M-F) characterized by severe bone-cartilage defects, subchondral cysts, and extensive osteophytes in the medial femoral compartment, which would render the determination of both the epicondylar axis and the AT location impossible radiologically. Advanced imaging techniques such as computed tomography (CT) or magnetic resonance imaging (MRI) can be used for these patients, but they are not practically useful and add additional time and cost. Therefore, for patients with Type M-F deformity who are candidates for total knee arthroplasty (TKA), a study will be conducted to determine the JL location observationally without interfering with the surgical technique, using both preoperative radiological measurements and intraoperative caliper measurements. The measurements will be repeated in postoperative X-rays, and the functional short-term outcomes will be evaluated over a period of two years.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years of age
* Candidates with varus alignment osteoarthritis of the knee
* Patients with complete data set
* Patients who have agreed to participate in the study

Exclusion Criteria:

* Patients who did not provide consent to participate in the study
* Patients with post-traumatic osteoarthritis
* Patients with inflammatory type of osteoarthritis
* Patients with incomplete data set

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with KL Grade 4 severe OA with type M severe varus malalignment or just KL4 OA with intraarticular type 3 and 4 deformity according to Parvizi classification of varus gonarthrosis
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Determination of joint Line according to adductor ratio | comparison between baseline (preoperative and intraoperative) measurements
  Comparison of preoperative and intraoperative measurement of Adductor ratio (adductor tubercle to joint line/transepicondylar width; mm/mm)

SECONDARY OUTCOMES:
Determination of joint Line according to distance from medial and lateral epicondyles to joint line | comparison between baseline (preoperative and intraoperative) measurements
  Comparison of preoperative and intraoperative measurements (mm)
HSS (Hospital for Special Surgery) knee score | comparison between preoperative and postoperative 12th month control
  The score evaluates a range of factors, and each factor is assigned a score on the 100-point scale and and higher scores indicate better functional status

CONTACTS AND LOCATIONS:
Overall Officials: murat altay, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Keçiören SUAM, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP